CLINICAL TRIAL: NCT01016158
Title: Umbilical Cord Serum Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Kyung-Chul Yoon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-2009-11-135
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Recurrent Corneal Erosion
Keywords: Umbilical cord serum; Recurrent corneal erosion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord serum eyedrops (Experimental): patients with recurrent corneal erosions were treated with 20% umbilical cord serum eye drops 3 to 4 times a day in addition to artificial tears
  Interventions: Drug: Umbilical cord serum eyedrops

INTERVENTIONS:
Drug: Umbilical cord serum eyedrops — 20% umbilical cord serum eye drops 3 to 4 times a day

SUMMARY:
In the present study, the investigators investigated the efficacy of umbilical cord serum eye drops for the treatment of patients with recurrent corneal erosions. Group A were treated with 20% umbilical cord serum eye drops 3 to 4 times a day in addition to artificial tears, and group B were treated with artificial tears only. Ophthalmic examinations including visual acuity measurement and slit lamp biomicroscopy were performed before and every month after treatment. Recurrence was defined as the presence of clinical symptoms accompanied by epithelial defects in the cornea.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent corneal erosions

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

REFERENCES:
- [Result] Yoon KC, Im SK, Park YG, Jung YD, Yang SY, Choi J. Application of umbilical cord serum eyedrops for the treatment of dry eye syndrome. Cornea. 2006 Apr;25(3):268-72. doi: 10.1097/01.ico.0000183484.85636.b6. PMID 16633024
- [Result] del Castillo JM, de la Casa JM, Sardina RC, Fernandez RM, Feijoo JG, Gomez AC, Rodero MM, Sanchez JG. Treatment of recurrent corneal erosions using autologous serum. Cornea. 2002 Nov;21(8):781-3. doi: 10.1097/00003226-200211000-00010. PMID 12410036
- [Result] Yoon KC, You IC, Im SK, Jeong TS, Park YG, Choi J. Application of umbilical cord serum eyedrops for the treatment of neurotrophic keratitis. Ophthalmology. 2007 Sep;114(9):1637-42. doi: 10.1016/j.ophtha.2006.12.014. Epub 2007 Mar 26. PMID 17382396